CLINICAL TRIAL: NCT06559631
Title: Adaptation of Community Reinforcement Approach for the Treatment of Drug Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Saghir (Other)
Responsible Party: Sponsor-Investigator, Muhammad Saghir, Director of clinical affaires, Clinical Psychologist, Principal Investigator, at Islamabad Rehab Clinic., International Islamic University, Islamabad
Organization: International Islamic University, Islamabad (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Adaptation of CRA
Record Dates: First submitted 2024-01-31; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Substance Use Disorders; Comorbidities and Coexisting Conditions
Keywords: Substance Use Disorders; Treatment Model; Comorbid Mental Disorders; Residential Treatment
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Research design of the study shall consists two-arms, single-blind randomized controlled trial (RCT). While Randomized Control Trial (RCT) shall consists of two groups: Active Treatment (AT) group and Control group
Who Masked: Participant, Outcomes Assessor
Masking Description: single-blind randomized controlled trial (RCT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Experimental group will receive the indigenously adapted Community Reinforcement Approach based psychotherapeutic sessions after the completion of drugs related detoxification (after 21 days since hospitalization) for 90-120 days in residential treatment.
  Interventions: Behavioral: Indigenously Adapted CRA
- Control Group: Treatment as usual (No Intervention): This group will receive treatment as usual which includes detoxification of drugs, general counselling for drug addiction prevention, 12 steps program and life skills training. Duration of residential treatment is between 90-120 days.

INTERVENTIONS:
Behavioral: Indigenously Adapted CRA — Treatment group will receive psychotherapy based on CRA which is an evidence based approach. This adapted version of CRA also consists emotional management, behavioral interventions, drug addiction treatment and islamically integrated psychotherapy for drug addiction and comorbid mental disorders.
  Arms: Treatment Group

SUMMARY:
Central idea of the study is to adapt a treatment program for drug addiction treatment indigenously and relapse prevention, and to establish its efficacy.

This study helps the society to have an evidence-based approach with proven efficacy to deal with drugs related issues in Pakistan along with minimizing the rate of relapse which is the major issue with current disease model for treatment of addiction in different rehabs within the country.

Present study's aim is to adapt culturally and islamically a robust treatment protocol: Reinforcement Approach (CRA) through randomized control trial to determine its efficacy in the field of drug addiction rehabilitation. Moreover, CRA is also be used with comorbid psychological illnesses. Because, in the treatment facilities disease model is currently prevailing which lacks empirical evidence, and they do not have proven efficacy.

DETAILED DESCRIPTION:
In this study CRA is adapted and prepared as a protocol for residential treatment for drug addiction and drug induced psychosis as well. Intervention is applied to patients admitted to Islamabad Rehab Clinic (IRC). 90 days treatment plan is developed based on CRA interventions along with religious interventions. These religious interventions are based on Islamically Integrated psychotherapy. After discharge from the treatment every participant will be monitored for next 3 months through follow up session with patient and caregivers as well.

In CRA, face to face interaction is required for intervention including 8 sessions for focuses on the reality of client's social environment so that for learning real life opportunities could be focused as per client needs to enhance engagement and learning.

For internal motivation and involvement in CRA, adaptations were added to enhance CRA's effectiveness. There were two major adaptations in CRA to make it accord with the cultural relevant with the targeted population. First adaptation is based on religion Islam. It includes several sections, and these sections are adapted in CRA's counseling goals. In first section morality is being adapted with CRA, morality is about the Islamically integrated ways about hygiene, sleep, eating, clothes, meeting others, physical health, happiness and sadness related. Second section is related to internal framework of human psyche, which comprises of Cognition (Aql), Behavioral inclination (Nafs), Sprit (Ruh), Emotion (Ihsaas) and Heart (Qalb). In third section principle of change and tazkia e nafs. There are three stages in principle of change: 1.Inkishaf, 2. Itidal and 3. Itehad.

Second adaptation is about the effective coping skills related therapeutic intervention, which is comprises of four distinctive categories such as emotional management, interpersonal effectiveness: assertiveness, habit formation and relapse prevention counseling.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted for treatment of drug addiction with or without comorbid psychological disorders.

Exclusion Criteria:

* Patient with no history of drug abuse.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Recovery | First assessment will be conducted at the time of admission which will be completed till 21 days after admission. Second assessment after 120 days at the time of discharge. Third outcome measure during the follow up at the sixth month after discharge.
  Staying in abstinence from the drug of abuse. Recovery will be measured through Addiction Recovery Questionnaire (ARQ), this is a 4 point rating scale which measures normal living, abstinence and positive expectancy as recovery's subscales.

SECONDARY OUTCOMES:
Comorbidities | First assessment will be conducted at the time of admission which will be completed till 21 days after admission. Second assessment after 120 days at the time of discharge. Third outcome measure during the follow up at the sixth month after discharge.
  comorbidities associated with substance use disorders will also be included and measured through Symptoms checklist-90 (SCL-90), 5 point rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mazhar Iqbal Bhatti, Study Chair — International Islamic University, Islamabad
Locations (2):
- Pakistan (2):
  - Hayat Rehab Clinic (HRC), Islamabad
  - Islamabad Rehab Clinic (IRC), Islamabad

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- See also: this is the link of a cite facility, Islamabad Rehab Clinic — https://ircl.pk/
- See also: this is the link of a cite facility, Hayat Rehab Clinic — https://hrci.pk/

DOCUMENTS (3):
  • Study Protocol (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT06559631/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT06559631/SAP_001.pdf
  • Informed Consent Form (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT06559631/ICF_002.pdf